CLINICAL TRIAL: NCT05045053
Title: Efficacy of Xiidra in the Management Dry Eye Disease After Corneal Collagen Cross Linking
Brief Title: Efficacy of Xiidra in Dry Eye Disease After Collagen Cross Linking
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, assisatant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hamaky17
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Corneal Disease
Keywords: dry eye; cross linking; xiidra
MeSH Terms: conditions — Corneal Diseases; Dry Eye Syndromes | interventions — lifitegrast; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant
Masking Description: computer based masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- xiidra group (Experimental): patients are treated with 0.5 % xiidra twice daily and artificial tears for 6 months after corneal collagen cross linking
  Interventions: Drug: Xiidra 5% Ophthalmic Solution
- control group (No Intervention): patient are treated with artificial tears for 6 months after corneal collagen cross linking in both groups

INTERVENTIONS:
Drug: Xiidra 5% Ophthalmic Solution — lifitegrast 0.5% ia applied twice daily after corneal collagen cross linking
  Other Names: lifitegrast
  Arms: xiidra group

SUMMARY:
dry eye disease after corneal collagen cross linking affect ocular function leading to reduced vision, photophobia, glare, halos, and foreign body sensation.

DETAILED DESCRIPTION:
first group of patients were treated with 0.5 % xiidra twice daily and artificial tears for 6 months.Second group treated with artificial tears for 6 months. the treatment starts after corneal collagen cross linking in both groups ,Baseline and post-treatment full ophthalmic examination was done.

ELIGIBILITY:
Inclusion Criteria:

* corneal collagen cross linking

Exclusion Criteria:

* systemic or ocular diseases ,previous ocular surgery, corneal pathology and contact lens wearers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change in Break up Time | 6 months
  fluorescein sodium stripes will be used for measurement of Break up Time in seconds at baseline and during the study

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Elhamaky, Principal Investigator — Benha university faculty of medicine
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates